CLINICAL TRIAL: NCT05871138
Title: Prognostic Value of Delta LUS Score of Patients Hospitalized for Acute Heart Failure Within 30 Days of Discharge
Brief Title: Prognostic Value of Delta LUS Score of Patients Hospitalized for Acute Heart Failure
Acronym: Deltalus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, clinical proffesor, University of Monastir
Other Study IDs: Delta- LUS
Record Dates: First submitted 2023-03-17; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Emergencies; Acute Heart Failure
Keywords: Delta-lus score; heart failure
MeSH Terms: conditions — Emergencies; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
prognostic value of delta LUS score of patients hospitalized for acute heart failure within 30 days of discharge.

DETAILED DESCRIPTION:
The aim of our study is to evaluate the contribution of the variation of the LUS score performed at the time of admission (LUS1) and at discharge (LUS2) in predicting the clinical course of patients admitted for acute cardiac decompensation 30 days after discharge.

Delta LUS score=((LUS2-LUS1) *100)/LUS1

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years,
* Patients hospitalized in the emergency department for dyspnea having as etiology an acute heart failure and in whom will be performed two pulmonary ultrasound examinations (at entry and exit).

Exclusion Criteria:

* Age less than 18 years
* Dyspnea of non-cardiac etiology (cause: pulmonary, traumatic, toxic...)
* Altered state of consciousness (Glasgow score<14)
* Hemodynamic instability: presence of peripheral signs of shock, use of vasoactive drugs
* Mechanical ventilation from the outset
* Cardiorespiratory arrest
* Inability to give consent to the study
* Missing one of two ultrasound examinations
* Unable to make telephone contact after one month.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study that will be conducted in the emergency department of CHU Fattouma Bourguiba Monastir over a period from March 2023 to December 2023.
  Will be included in this study patients aged over 18 years, hospitalized in the emergency department for dyspnea having as etiology an acute heart failure and in whom will be performed two pulmonary ultrasound examinations (at entry and exit). These patients will be contacted after one month of their discharge from the hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Delta lus | 30 days
  The primary outcome evaluate the contribution of the variation of the LUS score performed at the time of admission (LUS1) and at discharge (LUS2) in predicting the clinical course of patients admitted for acute cardiac
Readmission | 30 days
  Readmission

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Pr, Principal Investigator — University of Monastir
Locations (2):
- Tunisia (2):
  - Semir Nouira, Monastir, Monastur
  - Emergency Departement, Monastir